CLINICAL TRIAL: NCT05957991
Title: Danish Precocious Puberty Study (DAPP Study) A National Cohort Study on Incidence and Etiologies for Precocious Puberty
Brief Title: Danish Precocious Puberty Study - DAPP Study A National Cohort Study on Incidence and Etiologies for Precocious Puberty
Acronym: DAPP
Status: Not yet recruiting | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Rikke Beck Jensen, Associate Professor PhD, Copenhagen University Hospital at Herlev
Other Study IDs: DanishPrecociousPubertyStudy
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Puberty, Precocious
Keywords: Puberty
MeSH Terms: conditions — Puberty, Precocious | interventions — Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood sample for hormone analysis, genetic and epigenetic analysis Urine sample analysis of endocrine disrupting chemicals
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Met -lifestyle intervention: Girls with overweight and early puberty aged 8-9 years Treatment with metformin without lifestyle intervention (diet, training)
  Interventions: Drug: Metformin Hydrochloride tablet; Behavioral: No lifestyle intervention
- Met + lifestyle intervention: Girls with overweight and early puberty aged 8-9 years Treatment with metformin with lifestyle intervention (diet, training)
  Interventions: Drug: Metformin Hydrochloride tablet; Behavioral: Lifestyle intervention
- Placebo-lifestyle intervention: Girls with overweight and early puberty aged 8-9 years Treatment with placebo without lifestyle intervention (diet, training)
  Interventions: Drug: Placebo; Behavioral: No lifestyle intervention
- Placebo+lifestyle intervention: Girls with overweight and early puberty aged 8-9 years Treatment with placebo with lifestyle intervention (diet, training)
  Interventions: Drug: Placebo; Behavioral: Lifestyle intervention

INTERVENTIONS:
Drug: Metformin Hydrochloride tablet — Treatment with metformin
  Other Names: Metformin
  Groups: Met + lifestyle intervention; Met -lifestyle intervention
Drug: Placebo — Treatment with placebo
  Groups: Placebo+lifestyle intervention; Placebo-lifestyle intervention
Behavioral: Lifestyle intervention — Changing behaviour on diet and excersise
  Groups: Met + lifestyle intervention; Placebo+lifestyle intervention
Behavioral: No lifestyle intervention — No changes in behaviou on diet and excersise
  Groups: Met -lifestyle intervention; Placebo-lifestyle intervention

SUMMARY:
There is an urgent need to obtain more knowledge about the influence of weight and metabolism on the timing and progression of puberty. The age of pubertal onset has been constantly declining during the last decades and extremely early maturation may have yet unseen consequences for the psychosocial development of the child as well as detrimental long-term health consequences. Studies have shown that girls with early-onset puberty are more likely than their peers to enter sexual relationships at a younger age, to experience more psychological distress, and to engage in risk-taking behaviors. In addition, early maturation may have long-term health consequences since earlier menarche is associated with an increased risk of all-cause mortality and cardiovascular disease later in life in large epidemiological studies. The exact aetiology for the earlier onset of puberty in the general population remains to be elucidated, and the cause is probably to be found in a complex interplay between genetic, epigenetic, environmental and metabolic factors. However, world-wide there is a concerning increasing prevalence of overweight in childhood and early puberty is one of many consequences of this. Environmental factors such as endocrine disrupting chemicals have been suggested to play a role for both obesity and precocious puberty either directly or through epigenetic moderation. The current study of a Danish National cohort will explore the incidence and aetiology of precocious puberty for better treatment and prevention. Furthermore, a placebo-controlled randomized controlled trial may give a novel mechanistic insight of the interplay between insulin sensitivity and sex steroids. To our knowledge this study is the first of its kind and may lead to novel alternative treatment strategy for overweight girls with early puberty that may have beneficial effects on long-term morbidity and mortality.

DETAILED DESCRIPTION:
Original title of the project: Danish Precocious Puberty Study (DAPP study)

Project leaders and trial site: Principal investigator: Rikke Beck Jensen, MD PhD DMSc, Department of Children and Adolescents - Herlev Hospital Borgmester Ib Juuls Vej 101, 2730 Herlev, Denmark

Trial Site: 17 pediatric departments in Denmark

Purpose of the study: The development of precocious puberty is a growing problem worldwide. Breast development is observed as early as preschool age, which can have serious consequences for girls' quality of life. Previous studies have also found a correlation between early puberty and increased risk of diseases later in life. Lifestyle factors causing obesity have been suggested as a cause for the declining age of pubertal onset. Endocrine disrupting chemicals in our environment likely play a role as well. The purpose of this study is to determine the incidence of children experiencing early puberty in Denmark and to investigate the factors influencing the timing of pubertal onset. Our hypothesis is that environmental factors such as lifestyle and exposure to endocrine disrupting chemicals may affect pubertal onset either directly or through epigenetic changes.

Method, design and research procedures: The project is a national cohort study that will take place at 17 pediatric departments in Denmark. We will include all children referred with precocious puberty to the country's pediatric departments over a period of 3 years (September 2023-May 2026). We will examine the number of children referred with precocious puberty and investigate their BMI, metabolic function, levels of endocrine disrupting chemicals, as well as the genetic and epigenetic patterns. All examinations will be conducted at the 17 pediatric departments by doctors or nurses experienced in working with children. The study includes a clinical examination with pubertal assessment. Additionally, the children's growth will be assessed by measuring height, weight, hip-waist ratio, and blood pressure.

The clinical examination is supplemented by urine collection (approximately 50 ml) and blood sampling (approximately 35 ml). In the blood sample analyses of hormones, growth factors, markers for glucose metabolism, and blood lipids will be performed. The content of various endocrine disrupting chemicals such as phthalates and pesticides is determined in the urine.

DNA is isolated from the blood for investigation of genetic polymorphisms (single nucleotide polymorphisms, SNPs). We will focus on genes and variants with known or theoretical effects on hormone production and insulin sensitivity. Specific "primers" will be used for known SNPs or SNP arrays containing common variants found in more than 1% of the population. Methylation of DNA, known as epigenetics, will also be investigated. We will not examine hereditary diseases, and since we only examine known variants, no secondary findings will occur.

A questionnaire survey will be conducted as part of the study to map the children's early growth patterns, health, physical activity, as well as the growth and pubertal development of their parents. In addition, there are questions for both parents and children to determine the children's quality of life. The questionnaires are filled out online in REDCap, a secure web application for building and managing databases and online surveys.

Study participants: Approximately 1500 children will be recruited from the 17 pediatric departments in Denmark. This corresponds to the number of children expected to be referred to pediatric departments each year in a three year period based on previous registry data with clinical signs of early puberty.

Inclusion criteria: All children referred for suspected precocious puberty with one of the following ICD10 codes will be included: DE301, DE228A, DE308A, DE270B, DE308, DE309, DZ003. Patients with cancer or chronic diseases (e.g., previous malignant disease, chemotherapy, radiation, or known genetic disease) will also be included, even though these conditions themselves can affect pubertal onset. These patients are included to estimate the number of children with precocious puberty per year in Denmark.

Exclusion criteria: If we observe unexpected psychological or physical reactions or if participants are deemed unsuitable or withdraw their participation, they can be excluded at any time.

Recruitment of participants: The children will be recruited from all 17 pediatric departments, where they are referred by their general practitioners or school health nurses with signs of precocious puberty. All patients meeting the criteria for inclusion in the study will be invited to participate throughout the three-year inclusion period. Parents of potential participants will receive information about the study in their digital mailbox before their visit to the pediatric department, so they can bring a support person

Side effects, risks, and disadvantages: This research project involves no known health risks, side effects, or other burdens for the participants. However, some children may find the blood sampling procedure slightly uncomfortable, and they are offered a numbing patch to anesthetize the skin where the blood sample is taken. Pubertal assessment may be perceived as intrusive for some children, so all children will be examined by clinical staff experienced in pubertal assessment in children. Body composition will be assessed using bioimpedance, which can measure fat percentage in some of the pediatric departments. Children will not be exposed to radiation or radioactivity.

Financial considerations: Data collection for the study will be covered by a research grant from the Novo Nordisk Foundation totaling 9.89 million DKK. Expenses for blood and urine sample analyses will be covered by funds from private foundations. The study is not supported by the pharmaceutical industry, and there are no commercial interests associated with the study. Information about the financial support will be provided in the participant information material. Compensation for participation is not offered. No members of the project group have a specific affiliation with the funding sources, and the execution of this research project is solely controlled by the project leader, who has no financial interest in the research project's results.

ELIGIBILITY:
Inclusion Criteria:

• All children (> 4 years of age) referred to one of the seventeen collaborating pediatric departments with one of the following diagnosis (ICD10)

* DE301
* DE228A
* DE308A
* DE270B
* DE308
* DE309
* DZ003

Exclusion Criteria:

* If the investigating doctor at the local hospital observes unexpected psychological/physical reactions, or a participant is found to be unsuitable (cf. inclusion criteria) or regrets agreeing to participate, this person can at any given time be excluded.

Ages: 3 Years to 10 Years | Sex: All
Age Groups: Child
Study Population: Seventeen pediatric hospital departments in Denmark will be included and an expected more than 1,500 children referred for early puberty will be invited to participate in the study. Since this cohort consists of patients who are going through the examinations and blood samples as part of the routine clinical work-up for CPP we expect a high participation rate around 70-80%. The patients are asked for a fasting blood sample and a urine sample for the clinical biobank. It is essential to include all departments to evaluate the incidence of precocious puberty in Denmark and to ensure power for the analyses of etiology.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of CPP among all children referred to 18 Danish pediatric departments during a 3-year period | 3 years
  Number of patients referred who have precocious puberty
BMI (SDS) at pubertal onset | 3 years
  Adiposity in children with precocious puberty
Genome-wide methylation patterns in peripheral blood associated with CPP and treatment | 3 years
  epigenetic alterations
Urinary EDC excretion profiles in CPP children compared to age-matched controls | 3 years
  endocrine disrupting chemicals associated to early puberty
Randomised placebo controlled trial | 3 years
  The effect of metformin and/or lifestyle intervention on pubertal development

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (5):
  - Copenhagen University Hospital - Herlev, Herlev, Capital Region
  - Univerity Hospital Aalborg, Aalborg
  - University Hospital Aarhus, Aarhus
  - University Hospital Odense, Odense
  - University Hospital Roskilde, Roskilde

IPD SHARING:
Plan to Share IPD: Yes
Data collected in the study may be provided to qualified researchers with academic interest in precocious puberty. Shared data will be coded, with no protected health information included. Approval of the request are prerequisites to the sharing of data with the requesting party.
  Access to trial IPD can be requested by qualified researchers engaging in scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests may be submitted from 12 to 24 months after publication of the article.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA)